CLINICAL TRIAL: NCT00342212
Title: Actigraph Accelerometer Validation Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906131; 06-C-N131; NCT00602810 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Physical Activity
Keywords: Walking; Jogging; Bridging Study; Data Comparability; Healthy Adults; Healthy Volunteer; HV
MeSH Terms: conditions — Motor Activity

SUMMARY:
Background:

* Good measures of physical activity are needed for studies correlating physical activity and the risk of developing certain diseases.
* In preparation for use in a study of diseases and risk factors in Hispanic populations, NCI is evaluating a new model accelerometer to measure physical activity. An accelerometer is a small device worn on a belt at the waist that measures and records movement, capturing movement intensity and duration and associating it with clock-time.
* The new accelerometer (ActiGraph GTIM) uses a different type of motion detector from that used in the previous model (ActiGraph 7164).

Objective: To evaluate and compare the ActiGraph GTIM with the ActiGraph 7164 by collecting physical activity data using both models.

Eligibility: Men and women 18-74 years of age.

Design: Study participants wear both model accelerometers while they walk or jog around a track at several self-selected paces. Data from the two devices are compared.

DETAILED DESCRIPTION:
The NCI is collaborating with other NIH Institutes on a proposed extramurally funded longitudinal study of Hispanic subpopulations in the United States referred to as the Hispanic Community Health Study (HCHS). Hispanic populations are understudied with respect to many diseases and risk factors. To better understand the relationship between physical activity and chronic disease, and to make specific activity prescriptions, better methods are needed to improve the validity and reliability of physical activity assessment instruments to assess the frequency, duration, and intensity of physical activity. In preparation for use in the HCHS, NCI plans to evaluate a new type of accelerometer, a small device worn on a belt at the waist that measures and records movement, capturing movement intensity and duration and associating it with clock-time. This new accelerometer will be used in the HCHS to allow examination of levels as well as patterns of activity. Physical activity was measured with accelerometers in the nationally representative 2003-2006 National Health and Nutrition Examination Survey (NHANES). Between the time of the NHANES and the HCHS, there has been a change in the technology of the accelerometer used in NHANES. To allow comparison of the physical activity data that will be collected in the HCHS to the data collected with the previous technology used in NHANES, a cross-validation study is needed. The proposed study, the ActiGraph Accelerometer Validation Study, will compare the ActiGraph model 7164 used in NHANES with the new model GT1M to be used in the HCHS by simultaneously collecting physical activity data using both ActiGraphs under different circumstances of walking or jogging. The study will recruit 120 men and women ages 18-74, corresponding to the age range of the HCHS. Normal weight, overweight and obese participants will be included in each age/gender cell. Because the devices measure movement, it is not essential that the study participants be from any particular ethnic group. To derive comparable data for the 2 devices, the 2 accelerometer models will be worn on a belt, with one positioned on each hip. Study participants will be asked to walk/jog around a track for a known distance at several self-selected paces. Minute-by-minute and summary data from the two devices will be evaluated for comparability.

ELIGIBILITY:
* None given

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-03; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Westat, Inc., Rockville, Maryland
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Thomas S, Reading J, Shephard RJ. Revision of the Physical Activity Readiness Questionnaire (PAR-Q). Can J Sport Sci. 1992 Dec;17(4):338-45. PMID 1330274